CLINICAL TRIAL: NCT01530269
Title: C11-Sodium Acetate PET/CT Imaging for Metastatic Disease in Intermediate-to-high Risk Prostate Adenocarcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Phoenix Molecular Imaging (Other)
Responsible Party: Principal Investigator, Fabio Almeida MD, Medical Director and Principal Investigator, Phoenix Molecular Imaging
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: AMIC-AC-002
Record Dates: First submitted 2012-02-04; First posted 2012-02-09 (Estimated); Last update posted 2019-03-07 (Actual); Status verified 2019-03

CONDITIONS: Prostate Cancer; Prostate Adenocarcinoma
Keywords: intermediate; high; risk; radiation; therapy; planning; surgical; immunotherapy; chemotherapy; hormone
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Carbon-11

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- PET/CT imaging with C11-Sodium Acetate (Experimental)
  Interventions: Drug: C11-Sodium Acetate

INTERVENTIONS:
Drug: C11-Sodium Acetate — PET Imaging with C11-Sodium Acetate
  Other Names: C11 Acetate PET; Carbon 11; AC-PET

SUMMARY:
Positron emission tomography using carbon-11 acetate (AC-PET) may help find local or distant metastases from prostate cancer. This clinical trial is studying how this imaging test may help influence the choice and extent of initial treatments, and subsequent treatments.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the role of positron emission tomography using carbon-11 acetate (AC-PET) in the initial and subsequent management of patients with prostate cancer at intermediate or high risk for recurrence after initial curative therapy.
* Compare the value of AC-PET in predicting recurrence of prostate cancer with that of conventional approaches (e.g., pre-operative clinical staging, prostate-specific antigen, Gleason score, prostate and lymph node histology) in these patients.

ELIGIBILITY:
Inclusion Criteria:

Male patients will be studied who have prostate cancer:

* Diagnosed with prostate adenocarcinoma
* Has completed conventional staging examinations, including histologic evaluation with Gleason score, CT scan of the abdomen and pelvis, and whole-body bone scintigraphy Candidate for curative prostatectomy OR curative radiotherapy OR staging lymphadenectomy prior to surgery
* Deemed to be at intermediate or high risk for recurrence or metastatic disease after initial curative treatment, as defined by of one of the following:

  * Gleason score >= 7 or PSA >= 10
  * Gleason score < 7 or PSA <10 ng/mL with positive surgical margins, biopsy proven or suspected regional nodal involvement or conventional imaging showing limited metastatic disease that may be amenable to directed radiotherapy
  * Rising or non-responding PSA

Exclusion Criteria:

* < 18 years old
* claustrophobic patients

Ages: 18 Years to 90 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2012-04; Primary Completion 2019-01 (Actual); Study Completion 2019-01 (Actual)

PRIMARY OUTCOMES:
Tissue Biopsy of metastatic site(s) | Assessed within 30 days following AC-PET
  Patients will undergo needle biopsy of positive metastatic findings on C11- Acetate PET/CT

SECONDARY OUTCOMES:
PSA (prostate specific antigen) | Each 3 - 6 months for 24 months
  PSA (prostate specific antigen) will be monitored per routine clinical follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Fabio Almeida, MD, Principal Investigator — Medical Director, Phoenix Molecular Imaging
Locations (1):
- Phoenix Molecular Imaging, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: No